CLINICAL TRIAL: NCT05415202
Title: Remimazolam Safety and Efficacy for Nerve Blocks
Brief Title: Remimazolam Sedation for Nerve Blocks
Acronym: REMI-SEN
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jake Brandenburg, Assistant Professor, University of Utah
Other Study IDs: IRB_00149157
Record Dates: First submitted 2022-06-04; First posted 2022-06-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Procedural Anxiety; Procedural Pain
MeSH Terms: conditions — Pain, Procedural | interventions — remimazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Remimazolam Sedation: Patients receiving a nerve block prior to surgery or a re-block the day after surgery will receive remimazolam sedation for their nerve block.
  The nerve block will then be performed under standard conditions with standard monitors. Remimazolam will be used for sedation following the guidelines on the label.
  Dosing will be as follows:
  Induction of Procedural Sedation For adult patients: Administer 5 mg intravenously over a 1-minute time period. For ASA* III and IV patients: Administer 2.5 mg to 5 mg intravenously over 1 minute based on the general condition of the patient.
  Maintenance of Procedural Sedation (as needed) For adult patients: Administer 2.5 mg intravenously over 15 seconds. At least 2 minutes must elapse prior to administration of any supplemental dose.
  For ASA III and IV patients: Administer 1.25 mg to 2.5 mg intravenously over 15 seconds.
  At least 2 minutes must elapse prior to administration of any supplemental dose.
  Interventions: Drug: Remimazolam 20 MG [Byfavo]

INTERVENTIONS:
Drug: Remimazolam 20 MG [Byfavo] — Remimazolam will be administered for sedation and efficacy and safety will be recorded

SUMMARY:
Observational study recording sedation and safety of patients undergoing remimazolam sedation for peripheral nerve blocks.

Objectives:

To explore the safety and efficacy of remimazolam for neuraxial procedures and peripheral nerve pre-blocks and re-blocks.

Patients undergoing epidurals, fascial plane blocks, and peripheral nerve blocks will receive remimazolam for sedation.

Specific outcomes to assess include: depth of sedation, length of sedation, presence of apnea, presence of nausea/vomiting/other side effects, if the sedation was sufficient for the procedure.

Assessment methods:

MOAAS - Modified Observer's Assessment of Alertness and Sedation score Subjective patient report Vital signs Time for recovery Side effects

Hypothesis:

Remimazolam provides short-acting, adequate and safe sedation for peripheral nerve blocks in the ambulatory setting.

DETAILED DESCRIPTION:
Nerve blocks are short, mildly stimulating procedures that result in no increase in pain post-procedurally. They are often performed at our institution with sedation, typically midazolam with or without fentanyl.

Remimazolam is an intravenous sedative agent FDA approved for procedural sedation.

Remimazolam is an intravenous sedative agent FDA approved for procedural sedation. It has been shown to be safe and effective in outpatient colonoscopy and has demonstrated a faster recovery to neuropsychiatric function compared to midazolam.[i] It also has demonstrated decreased rates of hypotension and faster recovery time when compared to midazolam.i For high risk colonoscopies, similar rates of bradycardia and blood pressure changes have been found; and remimazolam was shown to be safe and short acting.[ii] For bronchoscopies, remimazolam continues to demonstrate faster return to neuropsychiatric function when compared to midazolam, as well as a safety profile equivalent to midazolam.[iii]

With a safety profile equivalent to midazolam but a much shorter duration of effect, it is a natural choice for a short, mildly stimulating procedures such as nerve blocks.

Patients will be identified by providers and study personnel according to inclusion and exclusion criteria by reviewing electronic charts of patients who will be receiving nerve blocks. Once identified as a possible pre-op block or re-block, then the patients will be approached and asked if they wish to participate in the study. Patient will be screened by chart review and questioning for allergies to remimazolam or dextran 40 and will be excluded if allergy is present.

After patients are identified by providers or study personnel as meeting the inclusion/exclusion criteria on the day of surgery, they will be approached and asked if they wish to participate in the study. If they choose to participate, then a provider or study personnel will perform the informed consent process.

BYFAVO (remimazolam) for injection is a benzodiazepine indicated for the induction and maintenance of procedural sedation in adults undergoing procedures lasting 30 minutes or less. For this study, remimazolam will be used according to its FDA approval, for procedural sedation in adults undergoing procedures lasting 30 minutes or less: peripheral nerve blocks, catheters, plane blocks, or epidural procedures. Route: Intravenous.

The nerve block will then be performed under standard conditions with standard monitors. Remimazolam will be used for sedation following the guidelines on the label.

Dosing will be as follows:

Induction of Procedural Sedation For adult patients: Administer 5 mg intravenously over a 1-minute time period. For ASA* III and IV patients: Administer 2.5 mg to 5 mg intravenously over 1 minute based on the general condition of the patient.

Maintenance of Procedural Sedation (as needed) For adult patients: Administer 2.5 mg intravenously over 15 seconds. At least 2 minutes must elapse prior to administration of any supplemental dose.

For ASA III and IV patients: Administer 1.25 mg to 2.5 mg intravenously over 15 seconds.

At least 2 minutes must elapse prior to administration of any supplemental dose.

MOASS scores will be assessed at baseline and frequently until 3 consecutive 5's are observed. The patient will be monitored until they have scored three consecutive 5's on the MOASS scale and their vital signs are stable. Any additional required sedative medications will be recorded, as will vital signs and side effects.

Supplemental oxygen may be administered as needed.

Patients are not eligible to participate in the study more than once.

[i] Rex, D. K., Bhandari, R., Desta, T., DeMicco, M. P., Schaeffer, C., Etzkorn, K., et al. (2018). A Phase III Study Evaluating the Efficacy and Safety of Remimazolam (CNS 7056) Compared with Placebo and Midazolam in Patients Undergoing Colonoscopy. Gastrointest. Endosc. 88 (3), 427-437.e6. doi:10.1016/j.gie.2018.04.2351

[ii] Rex, D. K., Bhandari, R., Lorch, D. G., Meyers, M., Schippers, F., and Bernstein, D. (2021). Safety and Efficacy of Remimazolam in High Risk Colonoscopy: A Randomized Trial. Dig. Liver Dis. 53 (1), 94-101. doi:10.1016/j.dld.2020.10.039

[iii] Pastis, N. J., Yarmus, L. B., Schippers, F., Ostroff, R., Chen, A., Akulian, J., et al. (2019). Safety and Efficacy of Remimazolam Compared with Placebo and Midazolam for Moderate Sedation during Bronchoscopy. Chest 155 (1), 137-146. doi:10.1016/j.chest.2018.09.015

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Will be receiving a pre-operative nerve block (single shot nerve block, nerve block catheter, plane block, epidural, etc.) or a re-block (a nerve block performed for pain control at least one day after surgery) from a qualified APS team member.

Exclusion Criteria:

1. Age less than 18 years.
2. Clinical instability or other condition preventing nerve block or sedation.
3. Pregnancy.
4. Inability to communicate quickly and efficiently their level of perceived sedation.
5. Allergy to remimazolam or dextran 40.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be identified by providers and study personnel according to inclusion and exclusion criteria by reviewing electronic charts of patients who will be receiving nerve blocks. Once identified as a possible pre-op block or re-block, then the patients will be approached and asked if they wish to participate in the study. Patient will be screened by chart review and questioning for allergies to remimazolam or dextran 40 and will be excluded if allergy is present.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change during procedure in Modified Observer's Assessment of Alertness/Sedation Scale score | Each minute during procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Sedation efficacy will be measured by serial scores on the Modified Observer's Assessment of Alertness/Sedation Scale (MOAAS: 5 is awake and alert, 0 is deep sedation). It will be measured each minute until 3 consecutive 5's are achieved.

SECONDARY OUTCOMES:
Nerve block completion or abortion | From just prior to initial remimazolam bolus at start of procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Will record if the nerve block was completed or aborted
Additional sedative requirement | From just prior to initial remimazolam bolus at start of procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Will record if additional sedative medications were required in order to achieve acceptable level of sedation in order to complete the procedure.
Oxygen Requirement | From just prior to initial remimazolam bolus at start of procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Oxygen requirement will be recorded. Will include liters per minute of oxygen administered as well as method of delivery.
Change in oxygen saturation as measured by pulse oximetry | From just prior to initial remimazolam bolus at start of procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Continuous pulse oximetry will be measured throughout the procedure and recorded every 2.5 minutes from prior to administration of remimazolam until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
Change in systolic blood pressure | From just prior to initial remimazolam bolus at start of procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Blood pressure will be measured and recorded every 2.5 minutes throughout the procedure from prior to initial administration of remimazolam until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
Change in diastolic blood pressure | From just prior to initial remimazolam bolus at start of procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Blood pressure will be measured and recorded every 2.5 minutes throughout the procedure from prior to initial administration of remimazolam until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
Change in mean arterial blood pressure | From just prior to initial remimazolam bolus at start of procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Blood pressure will be measured and recorded every 2.5 minutes throughout the procedure from prior to initial administration of remimazolam until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
Change in Heart Rate | From just prior to initial remimazolam bolus at start of procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Heart rate will be measured continuously and recorded every 2.5 minutes throughout the procedure from prior to initial administration of remimazolam until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
Required airway intervention | From just prior to initial remimazolam bolus at start of procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Any required airway intervention will be recorded including (but not limited to): intubation, mask ventilation, oral airway, positive pressure ventilation, reversal agent administration, procedure cancellation
Required hemodynamic intervention | From just prior to initial remimazolam bolus at start of procedure until 3 consecutive 5's on the MOAAS and at least 4 minutes from last administration of medication (up to 30 minutes)
  Any required hemodynamic intervention will be recorded including (but not limited to): reversal agent administration, vasoactive substance administration, procedure cancellation

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Brandenburg, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK, Bhandari R, Desta T, DeMicco MP, Schaeffer C, Etzkorn K, Barish CF, Pruitt R, Cash BD, Quirk D, Tiongco F, Sullivan S, Bernstein D. A phase III study evaluating the efficacy and safety of remimazolam (CNS 7056) compared with placebo and midazolam in patients undergoing colonoscopy. Gastrointest Endosc. 2018 Sep;88(3):427-437.e6. doi: 10.1016/j.gie.2018.04.2351. Epub 2018 Apr 30. PMID 29723512
- [Background] Rex DK, Bhandari R, Lorch DG, Meyers M, Schippers F, Bernstein D. Safety and efficacy of remimazolam in high risk colonoscopy: A randomized trial. Dig Liver Dis. 2021 Jan;53(1):94-101. doi: 10.1016/j.dld.2020.10.039. Epub 2020 Nov 23. PMID 33243567
- [Background] Pastis NJ, Yarmus LB, Schippers F, Ostroff R, Chen A, Akulian J, Wahidi M, Shojaee S, Tanner NT, Callahan SP, Feldman G, Lorch DG Jr, Ndukwu I, Pritchett MA, Silvestri GA; PAION Investigators. Safety and Efficacy of Remimazolam Compared With Placebo and Midazolam for Moderate Sedation During Bronchoscopy. Chest. 2019 Jan;155(1):137-146. doi: 10.1016/j.chest.2018.09.015. Epub 2018 Oct 4. PMID 30292760